CLINICAL TRIAL: NCT00006695
Title: BEAM Plus Iodine-131 Anti-B1 Antibody and Autologous Hematopoietic Stem Cell Transplantation for Treatment of Recurrent Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Brief Title: Monoclonal Antibody Therapy, Combination Chemotherapy, and Peripheral Stem Cell Transplant in Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0051-00-FB; COULTER-IND-3323 (Other Grant/Funding Number: Coulter Pharmaceuticals, Inc.)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Carmustine; Cytarabine; Etoposide; etoposide phosphate; Melphalan; Peripheral Blood Stem Cell Transplantation; tositumomab I-131

ARMS (1):
- Arm I (Experimental): Iodine-131 Anti-B1 Antibody/BEAM/autologous hematopoietic stem cell transplantation (AHSCT)
  Interventions: Drug: carmustine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: peripheral blood stem cell transplantation; Radiation: tositumomab and iodine I 131 tositumomab

INTERVENTIONS:
Drug: carmustine — 300 mg/m2 IV on Day -6
  Other Names: BCNU
Drug: cytarabine — 100 mg/m2 BID on Days -5 through -2
  Other Names: cytosine arabinoside
Drug: etoposide — 100 mg/m2 BID on Days -5 through -2
  Other Names: Etopophos, Toposar
Drug: melphalan — 140 mg/m2 IV on Day -1
  Other Names: Evomela
Procedure: peripheral blood stem cell transplantation — Following the chemotherapy, on Day 0 of treatment, the previously stored hematopoietic stem cells will be administered to the patient intravenously through a central line to the patient.
  Other Names: Autologous Hematopoietic Stem Cell Transplantation
Radiation: tositumomab and iodine I 131 tositumomab — Patients will receive two administrations of Iodine-131 Anti-B1 Antibody; the "dosimetric dose" and the "therapeutic dose". The dosimetric dose will consist of an infusion of unlabeled Anti-B1 Antibody (450 mg) immediately followed by an infusion of Anti-B1 Antibody (35 mg) which has been trace labeled with 5 mCi of Iodine-131 Anti-B1 Antibody. Using whole body anterior and posterior gamma camera scans and serial imaging studies over approximately one week, the clearance of the whole body dosimetric dose will be used to calculate the subsequent therapeutic dose of Iodine-131 Anti-B1 Antibody which delivers a total body dose of 75 cGy to the subject
  Other Names: Iodine-131 Anti-B1 Antibody

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well monoclonal antibody therapy, chemotherapy, and peripheral stem cell transplant work in treating patients with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rates and time to treatment failure in patients with relapsed or refractory non-Hodgkin's lymphoma treated with iodine I 131 monoclonal antibody anti-B1, followed by high-dose carmustine, etoposide, cytarabine, and melphalan (BEAM), and autologous peripheral blood stem cell transplantation (APBSCT) vs historical control patients treated with high-dose BEAM or carmustine, etoposide, cytarabine, and cyclophosphamide and APBSCT.
* Determine the safety of this regimen in these patients.

OUTLINE: Autologous peripheral blood stem cells (PBSC) are harvested and selected for CD34+ cells or granulocyte macrophage colony-forming units. On day -19, patients receive unlabeled monoclonal antibody anti-B1 (MOAB anti-B1) IV followed by a dosimetric dose of iodine I 131 MOAB anti-B1 IV over 20 minutes. On day -12, patients receive unlabeled MOAB anti-B1 IV followed by a therapeutic dose of iodine I 131 MOAB anti-B1 IV over 20 minutes. Patients then receive high-dose chemotherapy comprising carmustine IV on day -6, etoposide IV and cytarabine IV twice daily on days -5 to -2, and melphalan IV on day -1. Patients undergo autologous PBSC transplantation on day 0.

Patients are followed at days 30 and 100, at 6 months, and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-Hodgkin's lymphoma (NHL) of one of the following types:

  * Diffuse large B-cell
  * Composite (at least 50% of tumor showing diffuse histology)
  * Diffuse mixed cell
  * Immunoblastic
* Relapsed or refractory disease sensitive to initial or subsequent conventional therapy (at least a partial response)
* Eligible for high-dose carmustine, etoposide, cytarabine, and melphalan protocol and autologous bone marrow transplantation or peripheral blood stem cell transplantation
* Evidence of CD20 antigen expression in tumor tissue
* Bidimensionally measurable disease
* Adequate peripheral blood stem cells

  * At least 15,000,000 CD34+ cells/kg or
  * At least 25,000 granulocyte macrophage colony-forming units/kg
* Age: 19 to 70
* Performance status: Karnofsky 70-100%
* Life expectancy: at least 4 months post-transplantation
* Bilirubin less than 2.0 mg/dL
* Creatinine less than 2.0 mg/dL
* Cardiac ejection fraction at least 40% for any of the following criteria:

  * Age 60 and over
  * Significant cardiac history (myocardial infarction or congestive heart failure)
  * Received greater than 350 mg/m^2 of prior doxorubicin
* DLCO at least 50% of predicted
* HIV negative
* Fertile patients must use effective contraception during and for at least 6 months after study participation
* At least 4 weeks since prior biologic therapy and recovered
* Human antimouse antibody negative
* At least 4 weeks since prior cytotoxic chemotherapy and recovered
* At least 4 weeks since prior radiotherapy and recovered
* At least 4 weeks since prior immunosuppressants and recovered

Exclusion Criteria:

* No progressive disease in a field that has been previously irradiated with more than 3,500 cGy within the past year
* No known brain or leptomeningeal metastases
* No active obstructive hydronephrosis
* No New York Heart Association class III or IV heart disease
* No evidence of severe organ dysfunction
* No other major medical illnesses
* No active infection requiring IV antibiotics
* No other malignancy within the past 5 years except adequately treated skin cancer or carcinoma in situ of the cervix
* Not pregnant/negative pregnancy test
* No prior peripheral blood stem cell transplantation following high-dose chemotherapy or chemoradiotherapy
* No other concurrent biologic therapy for NHL
* No concurrent steroids except maintenance-dose steroids for noncancerous disease
* No concurrent external beam radiotherapy for NHL
* No other concurrent participation on protocol involving non-FDA-approved drugs or biologics

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2000-04-01 (Actual); Primary Completion 2005-09-01 (Actual); Study Completion 2014-12-16 (Actual)

PRIMARY OUTCOMES:
Event free survival rate | 100 days post transplant and at yearly intervals
  Participant survival without adverse events or progression

SECONDARY OUTCOMES:
Time to treatment failure | time of registration to time of treatment discontinuation or withdrawal for progression
  Time from registration to time of treatment discontinuation or withdrawal for progression
Overall survival | Time from registration to last participant death
  Time from first participant enrollment to last participant death or end of study

CONTACTS AND LOCATIONS:
Overall Officials: Julie M. Vose, MD, Study Chair — University of Nebraska
Locations (1):
- UNMC Eppley Cancer Center at University of Nebraska Medical Center, Omaha, Nebraska, United States